CLINICAL TRIAL: NCT06339892
Title: Comparison of Two Strategies for Monitoring HCMV Breakthrough Infections During Letermovir Prophylaxis. a Multicenter, Randomized, Open-label Trial
Brief Title: HCMV Breakthrough Infections During Letermovir Prophylaxis
Acronym: CMVbreak
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: Ministero della Salute, Italy (Other)
Responsible Party: Principal Investigator, Daniele Lilleri, Medical staff, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-3.11/451
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-03

CONDITIONS: Cytomegalovirus Infections; Cytomegalovirus Viremia; Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study (Experimental): Patients will stop LTV shifting to GCV/VGCV/FOS pre-emptive therapy in case of positive HCMV DNA and subsequent confirmation of productive infection by detection of DNAse-resistant HCMV plasma DNAemia. However, for safety reasons, patients of the Study arm will stop LTV and shift to pre-emptive therapy in case of HCMV DNAemia >10,000 copies/ml whole blood in two consecutive samples, even if DNAse-resistant HCMV plasma DNAemia is negative.
  Interventions: Diagnostic Test: Determination of HCMV DNA in plasma after DNAse digestion.
- Control (Active Comparator): Patients will stop LTV shifting to GCV/VGCV/FOS pre-emptive therapy in case of positive HCMV DNAemia confirmed in two consecutive samples.
  Interventions: Diagnostic Test: Determination of HCMV DNA in blood or plasma.

INTERVENTIONS:
Diagnostic Test: Determination of HCMV DNA in plasma after DNAse digestion. — Plasma will be tested after DNAse digestion for quantification of virion-associated HCMV DNA (defined as true breakthrough HCMV productive infection).
  Arms: Study
Diagnostic Test: Determination of HCMV DNA in blood or plasma. — HCMV DNA will be determined in blood or plasma without DNAse digestion, as per current clinical practice.
  Arms: Control

SUMMARY:
The goal of this clinical trial is to compare two strategies to monitor human cytomegalovirus (HCMV) infections in transplanted patients receiving letermovir (LTV) as anti-HCMV prophylaxis.

HCMV infection after transplantation is diagnosed by detection of HCMV DNA in blood. However, due to the peculiar mechanism of action of LTV, most episodes of HCMV DNA detection are caused by release in the blood stream of non-infectious HCMV DNA.

In true episodes of productive infection, HCMV DNA in blood is present inside the virion and therefore is resistant to DNAse digestion. Conversely, when non-infectious free-floating HCMV DNA is released in the bloodstream, it will be degraded after treatment of plasma with DNAse and will not be detectable by real-time PCR assays.

Researchers will compare determination of HCMV DNA in blood with or without previous digestion of non-infectious free-floating DNA with DNAse.

In patients of the Control group HCMV DNA will be tested without DNAse digestion. If HCMV DNA is positive, patients will stop LTV prophylaxis and receive antiviral therapy with another drug.

In patients of the Study group HCMV DNA will be tested after DNAse digestion. Only if HCMV DNA is positive after DNAse digestion, patients will stop LTV prophylaxis and receive antiviral therapy with another drug.

The main aim of the study is to demonstrate that, by avoiding inappropriate antiviral therapy during LTV prophylaxis, transplant patients will suffer of lower antiviral-drug-related toxicity. A monitoring strategy able to identify true episodes of HCMV productive infection during LTV prophylaxis will lead to a lower rate of inappropriate antiviral therapy and drug-related toxicity without an increased risk of HCMV disease.

DETAILED DESCRIPTION:
Patients will be enrolled at the start of conditioning regimen, and all patients of both arms will receive LTV prophylaxis after transplantation until day 100, according to standard procedures. Patients will be randomized (1:1) in two arms in case of positive HCMV DNAemia and will follow two different diagnostic strategies to assess HCMV refractivity to LTV prophylaxis.

* In the Control arm, patients will stop LTV shifting to GCV/VGCV/FOS pre-emptive therapy in case of positive HCMV DNAemia confirmed in two consecutive samples.
* In the Study arm, patients will stop LTV shifting to GCV/VGCV/FOS pre-emptive therapy in case of positive HCMV DNA and subsequent confirmation of productive infection by detection of DNAse-resistant HCMV plasma DNAemia. However, for safety reasons, patients of the Study arm will stop LTV and shift to pre-emptive therapy in case of HCMV DNAemia >10,000 copies/ml whole blood in two consecutive samples, even if DNAse-resistant HCMV plasma DNAemia is negative.

GCV/VGCV/FOS pre-emptive therapy will be stopped in all cases after detection of a negative HCMV DNAemia (i.e. below detection level of the assay adopted) in two consecutive samples.

After the end of LTV prophylaxis, HCMV infection will be treated with pre-emptive therapy according to current procedures of each center.

The hypothesis is that in the Study arm, due to the lower use of antiviral drugs as preemptive therapy, a significant reduction of neutropenia, renal failure and/or alteration in plasma electrolytes will be observed without an increase of HCMV diseases.

Study definitions

* Positive HCMV DNAemia will be defined as HCMV DNAemia >1,500 copies/ml whole blood (or >150 copies/ml plasma) for high-risk patients and >3,000 copies/ml whole blood (or >300 copies/ml plasma) for low-risk patients.
* HCMV disease will be defined by clinical and laboratory examination. Both proven and probable HCMV disease will be considered.
* Neutrophil impairment will be defined as delay in neutrophil engraftment and neutropenia after full engraftment will be defined by Common Terminology Criteria for Adverse Events version 4 (see website link below). Patients with 1 value of ANC < 1000/mmc (grade >= 3) from full engraftment to day 100 will be considered to have neutropenia.
* Acute renal impairment will be defined by Common Terminology Criteria for Adverse Events version 4 defined as sCr >2.0 x baseline sCr (grade >= 2).
* High risk: having a related donor with at least one mismatch at one of the specified three HLA gene loci (HLA-A, B, or DR); having an unrelated donor with at least one mismatch at one of the specified four HLA gene loci (HLA-A, B, C, and DRB1); having a haploidentical donor; the use of umbilical cord blood as the stem-cell source; the use of ex vivo T-cell-depleted grafts; and having GVHD of grade 2 or greater that led to the use of prednisone (or its equivalent) at a dose of 1 mg or more per kilogram of body weight per day.
* Low risk: all the patients who did not meet the definition of being at high risk

Antiviral drug-related toxicity will be considered as neutrophil impairment or kidney injury occurring at least 5 days after start of preemptive antiviral therapy.

Sample collection

* Virological monitoring: EDTA-treated blood for HCMV DNA quantification will be collected weekly until day 100, then monthly until day 360 (unless otherwise indicated by patient's clinical conditions). In case of positive HCMV DNAemia, virological monitoring will be performed twice a week.
* Immunological monitoring: heparin-treated blood will be collected i at day 100, 180 and 360 for determination of HCMV-specific T-cells.
* Neutrophil count: blood will be collected at least weekly in EDTA-treated tubes for blood cell count determination according to standard local procedures of each center.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years.
* Allogeneic hematopoietic stem cell transplant.
* HCMV IgG seropositivity before transplant
* Written informed consent.
* LTV prophylaxis administration

Exclusion Criteria:

* Age <18 years.
* Inability to comply with the requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
- Proportion of patients with positive HCMV DNAemia developing antiviral drug-related toxicity. | Day 100
  Antiviral drug-related toxicity will be considered as neutrophil impairment or kidney injury. Patients who exit before day 100 for death, underlying disease relapse, or transplant rejection after detection of HCMV-positive DNAemia will be considered as failures and counted along with antiviral drug-related toxicities for the analysis of the primary end-point occurring at least 5 days after start of preemptive antiviral therapy

SECONDARY OUTCOMES:
Proportion of patients developing HCMV DNAemia during LTV prophylaxis. | Day 100
Proportion of patients developing HCMV disease within day 100 and between day 100 and 360 from transplant (key secondary endpoint) | Day 100 and day 360
Proportion of patients stopping LTV prophylaxis and shifting to GCV/VGCV/FOS therapy. | Day 100
Proportion of patients requiring GCV/VGCV/FOS therapy between day 100 and 360. | Day 360
Proportion of patients with persisting HCMV DNAemia. | Day 360
  Positive DNAemia persisting two weeks after the first positive HCMV DNAemia.
Proportion of patients developing neutropenia between day 100 and 360. | Day 360
Proportion of patients developing HCMV-specific T-cell response at day 100, 180, and 360. | Day 100, day 180 and day 360
Proportion of patients developing LTV-resistant HCMV strains. | Day 100
Cumulative incidence of acute or chronic GvHD. | Day 100 and day 360
Transplant related mortality (TRM), underlying disease relapse, and 1-year survival. | Day 360

CONTACTS AND LOCATIONS:
Overall Officials: Fausto Baldanti, MD, Principal Investigator — Fondazione IRCCS Policlinico San Matteo
Locations (8):
- Italy (8):
  - ASST-Spedali Civili, Brescia, BS
  - Fondazione IRCCS Policlinico San Matteo, Pavia, PV
  - ASST-Ospedale Papa Giovanni XXIII, Bergamo
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Grande Ospedale Metropolitano "Bianchi-Melacrino-Morelli", Reggio Calabria
  - AOU Policlinico Umberto I, Roma
  - Policlinico Universitario Agostino Gemelli, Roma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marty FM, Ljungman P, Chemaly RF, Maertens J, Dadwal SS, Duarte RF, Haider S, Ullmann AJ, Katayama Y, Brown J, Mullane KM, Boeckh M, Blumberg EA, Einsele H, Snydman DR, Kanda Y, DiNubile MJ, Teal VL, Wan H, Murata Y, Kartsonis NA, Leavitt RY, Badshah C. Letermovir Prophylaxis for Cytomegalovirus in Hematopoietic-Cell Transplantation. N Engl J Med. 2017 Dec 21;377(25):2433-2444. doi: 10.1056/NEJMoa1706640. Epub 2017 Dec 6. PMID 29211658
- [Background] Ljungman P, Boeckh M, Hirsch HH, Josephson F, Lundgren J, Nichols G, Pikis A, Razonable RR, Miller V, Griffiths PD; Disease Definitions Working Group of the Cytomegalovirus Drug Development Forum. Definitions of Cytomegalovirus Infection and Disease in Transplant Patients for Use in Clinical Trials. Clin Infect Dis. 2017 Jan 1;64(1):87-91. doi: 10.1093/cid/ciw668. Epub 2016 Sep 28. PMID 27682069
- See also: Common Terminology Criteria for Adverse Events (CTCAE) — https://ctep.cancer.gov/protocolDevelopment/electronic_applications/ctc.htm